CLINICAL TRIAL: NCT04749407
Title: Dynamic Biomarkers of Immune Microenvironment for Stage III Locally Advanced Unresectable Non-small-cell Lung Cancer
Brief Title: Biomarkers of Stage III Locally Advanced Unresectable Non-small-cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: HZCH-2021-02
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: stage III locally advanced unresectable non-small-cell lung cancer; circulating tumor DNA; peripheral blood mononuclear cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chemoradiotherapy
  Interventions: Genetic: biomarker detection

INTERVENTIONS:
Genetic: biomarker detection — PBMC and ctDNA analysis

SUMMARY:
This study aims to dynamically monitor the expression profile status of peripheral blood mononuclear cells (PBMC) and the changes in circulating tumor DNA (ctDNA) levels in patients with stage III locally advanced unresectable non-small-cell lung cancer(NSCLC) after concurrent chemoradiotherapy or sequential chemoradiotherapy, and to explore biomarkers related to the immune microenvironment and the optimal time point for immunotherapy after chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent prior to any study specific procedures
2. Male or female aged over 18 years and under 70 years
3. Patients must have histologically- or cytologically-documented NSCLC who present with locally advanced, unresectable (Stage III) disease (according to Version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology [IASLC Staging Manual in Thoracic Oncology]), and clinical evaluation is suitable for concurrent chemoradiotherapy or sequential chemoradiotherapy
4. With measurable lesions (according to RECIST 1.1 criteria, long diameter of tumor lesions is 10mm, short diameter of lymph node lesions is 15mm).
5. World Health Organization (WHO) Performance Status of 0~2
6. Life expectancy ≥6 months
7. Adequate organ and marrow function as defined below:

   Absolute neutrophil count >1.5 x 109/L (1500 per mm3) Platelets >90 x 109/L (90,000 per mm3) Haemoglobin ≥9.0 g/dL (5.59 mmol/L) Serum creatinine CL >50 mL/min by the Cockcroft-Gault formula Serum bilirubin ≤1.5 x upper limit of normal (ULN) Total bilirubin (TBIL) ≤ 1.5 x upper limit of normal (ULN) In patients with no liver metastasis: AST and ALT ≤2.5 x ULN In patients with liver metastasis: AST or ALT ≤5 x ULN Urinary protein <2+; If the urine protein is ≥2+, the 24-hour urine protein quantification must show the protein to be ≤1g
8. International standardized ratio of normal coagulation function, no active bleeding and thrombosis disease International standardized ratio INR≤1.5×ULN Partial thromboplastin time APTT≤1.5×ULN Prothrombin time Pt ≤1.5 UlN
9. For women of non-surgical sterilization or reproductive age, use of a medically approved contraceptive method (such as an intrauterine device, birth control pills, or condoms) during the study treatment period and within 3 months after the study treatment period; Women of reproductive age who are not surgically sterilized must be negative for serum or urine HCG within 7 days prior to study enrolment; And must be non-lactation; Male patients who are not surgically sterilized or of reproductive age need to agree to use a medically approved method of contraception with their spouse for the duration of the study treatment period and for three months after the end of the study treatment period
10. Patients volunteered to participate in this study with good compliance and cooperated with multiple blood sample collection and follow-up

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. With other uncontrollable malignancies
2. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody
3. With any active autoimmune disease or a history of primary immunodeficiency (such as the following, but not limited to: autoimmune hepatitis interstitial pneumonia, uveitis, enteritis, hepatitis, the pituitary gland inflammation, vasculitis, nephritis, thyroid function, thyroid function is reduced, always had thyroid surgery must be incorporated into; Subjects with vitiligo or asthma in complete remission during childhood were included without any intervention as adults)
4. Patients are taking immunosuppressive or systemic or absorbable topical hormone therapy for immunosuppressive purposes (dose >10mg/day prednisone or other hormone) and continued to be used within 2 weeks before enrolment
5. Patients with congenital or acquired immune deficiency, such as HIV infection, or active hepatitis (transaminase does not meet the reference, hepatitis B: HBV DNA≥104/ml; hepatitis C: HCV RNA≥103/ml); Chronic hepatitis B virus carriers, HBV DNA<2000 IU/ml(<104 copies /ml) and must receive antiviral therapy during the trial to be included in the study
6. Patients with ≥2 grade pneumonitis from prior chemoradiation therapy
7. History of psychotropic substance abuse, alcohol abuse or drug abuse
8. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
9. Any condition that, in the opinion of the investigator, would interfere with study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage III locally advanced unresectable Non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with immune efficacy | up to 2 years
  According to the biomarker detection before and after chemoradiotherapy to identify biomarkers related to the immune microenvironment, including the expression levels of NK cells, T cells, B cells and other immune cells reflected by PBMC, as well as the expression levels of ctDNA
Optimal time for immunotherapy | up to 2 years
  Changes in the expression levels of ctDNA and PBMC immune cells before and after chemoradiotherapy to find the optimal time point for immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China